CLINICAL TRIAL: NCT01857765
Title: How Rehabilitation Affects the Time to Pain-free Living After Endoscopic Transaxillary Subpectoral Breast Augmentation
Brief Title: Breast Augmentation Rehabilitation Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The resident in charge of the project has graduated so we decided to close this study
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H11-02077
Record Dates: First submitted 2013-05-09; First posted 2013-05-20 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Breast Implants; Surgery, Plastic
Keywords: rehabilitation; reconstructive surgery
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Follow-up
- Rehabilitation (Experimental)
  Interventions: Behavioral: Rehabilitation; Behavioral: Follow-up

INTERVENTIONS:
Behavioral: Rehabilitation — Range of motion stretching exercises
  Arms: Rehabilitation
Behavioral: Follow-up — Follow-up with surgeon's clinic

SUMMARY:
The purpose of this study is to determine whether implementing a rehabilitation program can improve the post-operative time to pain free living after breast augmentation.

ELIGIBILITY:
Inclusion Criteria:

* women who undergo endoscopic transaxillary subpectoral breast augmentation
* women above the age of 18 years
* women with a BMI 18-27

Exclusion Criteria:

* women who underwent previous breast reconstruction (cosmetic or therapeutic)
* women who underwent previous chest surgery
* women with previous chest trauma
* women who underwent previous shoulder/arm surgery
* women with previous shoulder/arm injury
* women who smoke
* women who are Immunocompromised

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Time to return to baseline as measured on Visual Analogue Scale for pain | Baseline, six months, and one year after surgery

SECONDARY OUTCOMES:
Time to return to bilateral shoulder baseline range of motion | Baseline, six months, and one year after surgery
Change in psychosocial outcomes as measured by the BREAST-Q questionnaire | Baseline, six months, and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erin Brown, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada